CLINICAL TRIAL: NCT05567016
Title: Child Health and Infection With Low Density (CHILD) Malaria, a Randomized Controlled Trial to Assess the Long-term Health and Socioeconomic Impact of Interventions Targeting Low-density Malaria Infection (LMI) Among Children in Tanzania
Brief Title: CHILD (Child Health and Infection With Low Density) Malaria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Ifakara Health Institute (Other); Swiss Tropical & Public Health Institute (Other); Stanford University (Other); Chan Zuckerberg Biohub (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DMID protocol 21-0046; U01AI155315 (NIH)
Record Dates: First submitted 2022-09-30; First posted 2022-10-05 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Malaria,Falciparum; Malaria
Keywords: malaria; child health; chronic infection; subclinical infection; patent infection; subpatent infection; active case detection; passive case detection; fever case management
MeSH Terms: conditions — Malaria, Falciparum; Malaria; Persistent Infection; Asymptomatic Infections | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Individual randomized controlled trial
Masking Description: This will be an open label randomized controlled trial. Participants and personnel administering the intervention will be unblinded. Assessment of the primary outcome will be unblinded. Assessment of several secondary outcomes will be blinded as feasible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active Case Detection using molecular testing (ACDm) (Experimental): Per standard of care, children will receive passive case detection (PCD) using rapid diagnostic test (RDT) if they present with fever.
  Children will receive malaria active case detection (ACD) using RDT and qPCR (quantitative polymerase chain reaction) three times yearly with treatment using artemether-lumefantrine (AL) if RDT or qPCR positive.
  Interventions: Other: Active case detection using molecular testing (ACDm)
- Passive Case Detection using molecular testing (PCDm) (Experimental): Children who present with fever will receive PCD using RDT and qPCR with treatment using AL if RDT or qPCR positive.
  Per standard of care, children will not receive malaria ACD.
  Interventions: Other: Passive case detection using molecular testing (PCDm)
- Standard passive case detection (PCD) (Active Comparator): Per standard of care, children will receive PCD using RDT.
  Per standard of care, children will not receive malaria ACD.
  Interventions: Other: Control (standard of care)

INTERVENTIONS:
Other: Active case detection using molecular testing (ACDm) — In the ACDm arm, children will receive ACD using RDT and qPCR 3x yearly with treatment using artemether-lumefantrine (AL) if RDT or qPCR positive. With fevers, participants will receive standard PCD using RDT.
  Arms: Active Case Detection using molecular testing (ACDm)
Other: Passive case detection using molecular testing (PCDm) — With fevers, participants will receive PCDm, in which qPCR will be done in RDT negatives with treatment using AL if positive.
  Arms: Passive Case Detection using molecular testing (PCDm)
Other: Control (standard of care) — With fevers, participants will receive standard PCD using RDT with treatment using AL if positive.
  Arms: Standard passive case detection (PCD)

SUMMARY:
This trial will assess the long-term health and socioeconomic impact of interventions targeting low-density malaria infection (LMI) among children in Tanzania

DETAILED DESCRIPTION:
This is a 3-arm open-label randomized control trial of 600 children aged 6 months to 10 years in Tanzania, where transmission is low and a high proportion of infections are low-density. Standard of care based on passive case detection (PCD) using rapid diagnostic test (control arm) will be compared to two different approaches to detect and treat P. falciparum LMI: active case detection using molecular testing (ACDm) and PCD using molecular testing (PCDm). Aims are:

1. To assess the impact of standard PCD plus ACDm vs standard PCD on long-term child health
2. To assess the impact of PCDm vs standard PCD on long-term child health
3. To evaluate the cost-effectiveness of ACDm and PCDm

ELIGIBILITY:
Inclusion Criteria:

1. 6 months to 10 years of age of age at enrollment
2. Primary residence in the study area during the study period
3. Agree to come to study clinic for any illness
4. Agree to avoid medications outside the study, even herbal medication

Exclusion Criteria:

1. Another child from household already randomly selected for recruitment
2. Not able or does not provide informed consent
3. Need for emergency intervention
4. Known history of chronic illness requiring regular specialty care including diabetes mellitus, cancer, or Stage 3 or 4 HIV/AIDS
5. Contraindications to artemether-lumefantrine (AL) including history of allergic reaction, weight under 5 kg
6. Participation in another active/ongoing intervention trial

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2023-07-18 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2025-11-28 (Actual)

PRIMARY OUTCOMES:
Incidence of all-cause sick visits | 24-30 months from enrollment
  Number of sick visits to health facility per person time, excluding planned admissions for medical care, elective surgery, and trauma.

SECONDARY OUTCOMES:
Prevalence of anemia | 24-30 months from enrollment
  Proportion of routine Hb measurements that are low (<11 g/dL) or moderate-severe low (<8 g/dL)
Prevalence of underweight status | 24-30 months from enrollment
  Prevalence of underweight status will be defined as the percentage of participants with low weight for age z-scores of less than -2. The World Health Organization (WHO) anthropometric indices will be utilized for standards.
Prevalence of stunting | 24-30 months from enrollment
  Prevalence of stunting will be defined as the percentage of participants with low height for age z-scores of less than -2. The World Health Organization (WHO) anthropometric indices will be utilized for standards.
Prevalence of wasting | 24-30 months from enrollment
  Prevalence of wasting will be defined as the percentage of participants with low weight for height z-scores of less than -2. The World Health Organization (WHO) anthropometric indices will be utilized for standards.
Prevalence of malnutrition | 24-30 months from enrollment
  Prevalence of malnutrition will be defined as the percentage of participants with a z-score of -3 to -2 indicating moderate malnutrition or a z-score of less than -3 indicating severe malnutrition in any of the following: weight for age, height for age, or weight for height.
Prevalence of vomiting following administration of study drugs | 24-30 months from enrollment
  Vomiting immediately or within 30minutes following administration of study drugs and measures of non-adherence.
All-cause fever episodes | 24-30 months from enrollment
  Number of fever episodes (reported fever in the past 48hrs and/or axillary temperature of ≥37.5°C) per person time
Incidence of clinical symptoms | 24-30 months from enrollment
  Number of days with overall symptoms reported as moderate (≥3 on a 5-point scale) per person time
Incidence of clinical malaria | 24-30 months from enrollment
  New episodes of positive malaria test (with fever or other clinical symptoms) per person time
Proportion of fever episodes with clinical failure | 24-30 months from enrollment
  Proportion of fever episodes that lead to clinical failure, defined as persistent or worsening symptoms assessed 7 and 28 days after initial evaluation.
Prevalence of parasitemia | 24-30 months from enrollment
  Proportion of routine samples with parasites detected by microscopy or quantitative polymerase chain reaction (qPCR).
Incidence in antibiotics prescribed | 24-30 months from enrollment
  Number of antibiotic regimens prescribed per person time
Cognitive ability among children 0-3.4 years of age on the Global Scales of Early Development (GSED) | 24-30 months from enrollment
  GSED is a validated instrument that measures population-level early childhood development. The tool measures children's early skills and behaviors in four primary domains: motor, cognitive, language, and social-emotional development.Measures will be normalized within our sample to mean 0 and standard deviation 1, with higher scores indicating better test performance.
Cognitive ability among children 3.5-5 years of age on the International Development and Early Learning Assessment (IDELA) | 24-30 months from enrollment
  The IDELA is a validated, global tool that uses direct child assessment to measure early learning and development across 4 core domains (Emergent Literacy, Emergent Numeracy, Motor, Social-emotional). Scores range from 0-100% as a percentage of correct tasks averaged across the 4 domains. Measures will be normalized within our sample to mean 0 and standard deviation 1, with higher scores indicating better test performance.
Cognitive ability among children 6-12 years of age on the East Africa Neurodevelopment Assessment Tool | 24-30 months from enrollment
  The East African Neurodevelopment Assessment Tool is a locally adapted modification of the Kaufman Brief Intelligence Test 2nd Ed. The test assesses 3 core metrics including general intelligence, executive function, literacy skills - in addition to behavioral and emotional development. Measures will be normalized within our sample to mean 0 and standard deviation 1, with higher scores indicating better test performance.
Sustained attention among children 5-8 years of age on the Pencil Tapping Test | 24-30 months from enrollment
  The pencil tapping test is one of the tasks in the Preschool Self-Regulation Assessment (PSRA) and is used to assess inhibitory control in younger children. The child and an assessor have pencils, and child is instructed to tap one/two times(s) depending on what assessor does, with the number of correct responses scored. Measures will be normalized within our sample to mean 0 and standard deviation 1, with higher scores indicating better test performance.
Sustained attention among children 9-12 years of age on the Code Transmission Test, a local adaptation of the Test of Everyday Attention for Children(TEA-Ch) | 24-30 months from enrollment
  Code transmission test is a sub-test of Test of Everyday Attention for Children (TEA-Ch) used for assessment of sustained attention in children. In the test, the child must remember spoken digits, and remember the digit that comes before sequence of numbers. Child is scored on completed and correct answers. Measures will be normalized within our sample to mean 0 and standard deviation 1, with higher scores indicating better test performance.
Incidence of school absenteeism | 24-30 months from enrollment
  The number of days of school absenteeism for any reason including illness.
School performance | 24-30 months from enrollment
  School performance will be defined as the incidence of school advancement to the next grade.
Socioeconomic costs to participant | 24-30 months from enrollment
  Estimated long-term income loss due to impaired early childhood development
Socioeconomic costs to family | 24-30 months from enrollment
  Total caregiver-reported costs of sick visits and transport to sick visits plus estimated loss of income from number of days of caregiver work absenteeism.
Socioeconomic costs to health system | 24-30 months from enrollment
  Estimated costs of testing and treatment for caregiver-reported number of sick visits.
Cost effectiveness | 24-30 months from enrollment
  Cost per outcome averted (e.g., per sick visit averted, per disability adjusted life years (DALYs), and per economic dollar saved, etc.)
Prevalence of systemic inflammation | 24-30 months from enrollment
  Proportion of sick visits with elevated elevated C-reactive pep-tide (CRP)
Proportion with antimalarial antibodies against P.falciparum | 24-30 months from enrollment
  Percentage of patients with antimalarial antibodies
Proportion with biomarkers of inflammation | 24-30 months from enrollment
  Percentage of patients with elevated cytokines
Proportion with general antibody responses to vaccines | 24-30 months from enrollment
  Percentage of patients with vaccine antibodies
Proportion with general antibody responses to common pathogens | 24-30 months from enrollment
  Percentage of patients with common pathogen antibodies
Incidence of adverse events (AEs) | 24-30 months from enrollment
  Number of AEs per person time. AEs will be considered as any grade 3-4 AE or serious adverse event (SAE); individual AEs; or AEs related to study drugs.
Incidence of wasting | 24-30 months from enrollment
  Incidence proportion of wasting will be defined for each age range of measurement. It is defined as the proportion of children not wasted at the start of the period who became wasted during the age period (the proportion of children who had the onset of new episodes during the period). Incident wasting episodes are defined as a change in weight-for-length z-scores from above -2 Z in the prior measurement to below -2 Z in the current measurement. We will define incident severe wasting analogously using a -3 Z cutoff. We will assume a 60-day washout period before a new wasting episode could occur.
Incidence of stunting | 24-30 months from enrollment
  Incidence proportion of stunting will be defined for each age range of measurement. It is defined as the proportion of children not stunted at the start of the period who became stunted during the age period. Incident stunting episodes will be defined as a change in length-for-age z-scores from above -2 Z in the prior measurement to below -2 Z in the current measurement. We will define incident severe stunting analogously using a -3 Z cutoff.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hsiang, MD, MSc, Principal Investigator — University of California, San Francisco; Ally Olotu, MD, PhD, Principal Investigator — Ifakara Health Institute
Locations (1):
- Kiwangwa and Fukayosi clinics, Bagamoyo, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Summary results information will be submitted to ClinicalTrials.gov within 12 months of completion of follow-up of all study participants. After completion of the clinical trial, un-blinding will be performed, and results will be disseminated widely by presentation at international scientific meetings, in reports and policy meetings for local, regional, and global stakeholders, and in publications in peer-reviewed journals. Upon completion of planned analyses and publication of the main trial results, data will be made available for research purposes to other individuals in the scientific community upon request to the PI and Consortium PIs. Informed consent documents for the study will include a specific statement relating to posting and sharing of study information at ClinicalTrials.gov, and in presentations, reports, and publications, and that no individual identities will ever be used in these materials and forums.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Upon completion of analysis and publication of main trial results
Access Criteria: Request and approval of PIs Planned analyses completed and main trial results published

REFERENCES:
- [Derived] Jebiwott S, Gutapaka N, Sumari D, Loss G, Athuman T, Nyandele JP, Cummins H, Chemba M, Benjamin-Chung J, Gangar P, Wu X, Smith J, Chen I, Dorsey G, Fink G, Olotu A, Hsiang M. Child Health and Infection with Low Density (CHILD) malaria: a protocol for a randomised controlled trial to assess the long-term health and socioeconomic impacts of testing and treating low-density malaria infection among children in Tanzania. BMJ Open. 2024 Mar 27;14(3):e082227. doi: 10.1136/bmjopen-2023-082227. PMID 38538037

DOCUMENTS (2):
  • Informed Consent Form: Parent/Guardian consent for minor (2025-04-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT05567016/ICF_000.pdf
  • Informed Consent Form: Assent form for minors (2025-04-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT05567016/ICF_001.pdf